CLINICAL TRIAL: NCT00002162
Title: A Randomized, Parallel Arm, Comparative, Open Label, Multicenter Study of the Activity and Safety of Two Formulations of Saquinavir in Combination With Other Antiretroviral Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229D; NV15355
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Saquinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Saquinavir; Lamivudine; Stavudine; Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Saquinavir
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To evaluate the antiviral activity and safety of two formulations of saquinavir in combination with licensed nucleoside antiretroviral drugs.

DETAILED DESCRIPTION:
Patients are randomized to receive either hard gel or soft gel capsules of saquinavir in combination with at least one licensed nucleoside antiretroviral. Treatment will continue for 48 weeks. After the first 16 weeks, patients will be given the opportunity to roll over to the saquinavir formulation of choice.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Antiretroviral naiveness (i.e., less than 4 weeks of prior treatment) to at least one of the licensed nucleoside drugs.
* No more than 2 weeks of prior treatment with a protease inhibitor.
* No active opportunistic infection or other serious AIDS-defining condition.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malabsorption or inadequate oral intake.
* Lab or clinical abnormality worse than grade 3 (other than exercise-induced CPK elevations).
* Unexplained, chronic diarrhea, defined as more than three loose stools per day persisting for 2 weeks or more within the month prior to study entry.
* Active malignancy or anticipated need for chemotherapy during the study.
* Anticipated need for disallowed medications during the study.

Concurrent Medication:

Excluded:

* Other protease inhibitors.

Prior Medication:

Excluded:

* More than 4 weeks of the prior nucleoside antiretroviral selected for the patient's regimen.
* More than 2 weeks of any protease inhibitor.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140

CONTACTS AND LOCATIONS:
Locations (27):
- United States (23):
  - Phoenix Body Positive, Phoenix, Arizona
  - UCLA AIDS Clinical Research Ctr / Dept of Medicine, Los Angeles, California
  - AIDS Research Ctr, Palo Alto, California
  - UCD Med Ctr, Sacramento, California
  - UCSD Treatment Ctr, San Diego, California
  - Mount Zion Hosp of UCSF, San Francisco, California
  - San Francisco Veterans Adm Med Cntr, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Saint Joseph's Hosp, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Tulane Univ / Tulane / LSU Clinical Trials Unit, New Orleans, Louisiana
  - New England Med Ctr, Boston, Massachusetts
  - Harvard Univ / Massachusetts Gen Hosp, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - St Vincents Hosp and Med Ctr / AIDS Cntr Progrm, New York, New York
  - Univ of Oklahoma, Oklahoma City, Oklahoma
  - Univ of Pennsylvania / Division of Infectious Disease, Philadelphia, Pennsylvania
  - Univ of Texas Med Branch, Galveston, Texas
  - Infectious Diseases Association of Houston, Houston, Texas
- Canada (4):
  - Southern Alberta HIV Clinic / Foot Hills Hosp, Calgary, Alberta
  - Saint Paul's Hosp / Canadian HIV Trials Network, Vancouver, British Columbia
  - McMaster Univ Med Ctr, Hamilton, Ontario
  - Montreal Gen Hosp / Div of Clin Immuno and Allergy, Montreal, Quebec

REFERENCES:
- [Background] Cadman J. Roche brings new formulation of saquinavir to FDA. Food and Drug Administration. GMHC Treat Issues. 1997 Apr-May;11(4/5):8. PMID 11364377
- [Background] Mitsuyasu RT, Skolnik PR, Cohen SR, Conway B, Gill MJ, Jensen PC, Pulvirenti JJ, Slater LN, Schooley RT, Thompson MA, Torres RA, Tsoukas CM. Activity of the soft gelatin formulation of saquinavir in combination therapy in antiretroviral-naive patients. NV15355 Study Team. AIDS. 1998 Jul 30;12(11):F103-9. doi: 10.1097/00002030-199811000-00001. PMID 9708399